CLINICAL TRIAL: NCT01859429
Title: Stepped Care - Optimising Psycho-oncological Care Provision by Structured Screening and Diagnosis
Acronym: STEPPEDCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Susanne Singer, Susanne Singer, Prof. PhD MSc Epidemiology, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NKP-332-026
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Cancer
Keywords: Cancer patients; Psycho-oncological Care Provision; Structured Screening; Stepped care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepped Care (Experimental): Structured stepped requirement of psychosocial support
  Interventions: Other: Stepped Care
- Care as usual (No Intervention): Unstructured requirement of psychosocial support

INTERVENTIONS:
Other: Stepped Care — Step 1: Screening for psychosocial distress Step 2: If a patient is moderately or highly distressed according to step 1, the physician performs a brief structured interview and arranges, if necessary, appropriate psychosocial care Step 3: psychosocial care as indicated by step 2
  Arms: Stepped Care

SUMMARY:
The study will examine whether the provision of psychosocial support services for cancer patients in acute care can be optimized by the use of a structured combination of screening procedures with physician interviews and structured patient pathways.

There is strong evidence that a third of all cancer patients in acute care are suffering from mental health conditions and that a third expresses the need for professional psycho-oncological support.

However, physicians and nurses do not always identify these patients in need for support. Screening questionnaires are significantly better to identify distressed patients however the use of screenings alone does not necessarily improve the patients' emotional well-being.

Purpose of this study is to evaluate a psychosocial stepped care model which aims to decrease the patients' distress.

ELIGIBILITY:
Inclusion Criteria:

* patients in acute care for cancer
* written informed consent
* 18 years and older
* ability to complete questionnaires

Exclusion Criteria:

- insufficient command of German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mental condition | from baseline until 6 months
  Hospital Anxiety and Depression Scale, HADS

SECONDARY OUTCOMES:
Social functioning | from baseline until 6 months
  Role Functioning Subscale, EORTC QLQ-C30
Satisfaction with treatment | at discharge from acute care hospital, 6 months after admission to acute care hospital
  Quality of Care from the Patients Perspective, QPP
Comorbid mental disorders | at discharge from acute care hospital, 6 months after admission to acute care hospital
  Structured Clinical Interview for DSM-IV, SCID
Use of healthcare services | 6 months after admission to acute care hospital
  Questionnaire from the German Federal Health Survey (Bundesgesundheitssurvey)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Singer, PhD, Principal Investigator — Johannes Gutenberg University of Mainz
Locations (1):
- University of Leipzig, Dept. Psychosomatic Medicine and Psychotherapy, Leipzig, Germany

REFERENCES:
- [Background] Singer S, Danker H, Briest S, Dietrich A, Dietz A, Einenkel J, Papsdorf K, Lordick F, Meixensberger J, Mossner J, Niederwieser D, Prietzel T, Schiefke F, Stolzenburg JU, Wirtz H, Kersting A. Effect of a structured psycho-oncological screening and treatment model on mental health in cancer patients (STEPPED CARE): study protocol for a cluster randomized controlled trial. Trials. 2014 Dec 10;15:482. doi: 10.1186/1745-6215-15-482. PMID 25491069
- [Background] Singer S, Danker H, Roick J, Einenkel J, Briest S, Spieker H, Dietz A, Hoffmann I, Papsdorf K, Meixensberger J, Mossner J, Schiefke F, Dietel A, Wirtz H, Niederwieser D, Berg T, Kersting A. Effects of stepped psychooncological care on referral to psychosocial services and emotional well-being in cancer patients: A cluster-randomized phase III trial. Psychooncology. 2017 Oct;26(10):1675-1683. doi: 10.1002/pon.4492. Epub 2017 Jul 20. PMID 28665542
- [Background] Singer S, Roick J, Meixensberger J, Schiefke F, Briest S, Dietz A, Papsdorf K, Mossner J, Berg T, Stolzenburg JU, Niederwieser D, Keller A, Kersting A, Danker H. The effects of multi-disciplinary psycho-social care on socio-economic problems in cancer patients: a cluster-randomized trial. Support Care Cancer. 2018 Jun;26(6):1851-1859. doi: 10.1007/s00520-017-4024-x. Epub 2017 Dec 21. PMID 29270828
- [Derived] Singer S, Danker H, Meixensberger J, Briest S, Dietz A, Kortmann RD, Stolzenburg JU, Kersting A, Roick J. Structured multi-disciplinary psychosocial care for cancer patients and the perceived quality of care from the patient perspective: a cluster-randomized trial. J Cancer Res Clin Oncol. 2019 Nov;145(11):2845-2854. doi: 10.1007/s00432-019-03018-7. Epub 2019 Sep 10. PMID 31506739